CLINICAL TRIAL: NCT01596374
Title: Clinical Relevance of ROS (V-ros UR2 Sarcoma Virus Oncogene Homolog) Aberrations in Solid Tumours
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/01714
Record Dates: First submitted 2012-04-02; First posted 2012-05-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Alterations involving the ROS (v-ros UR2 sarcoma virus oncogene homolog 1) gene such as mutations, overexpression and gene rearrangements has been implicated in carcinogenesis and has been demonstrated to be a relevant target for ALK inhibitors. While emerging reports have demonstrated the role of ROS rearrangement in non-small cell lung cancer and cholangiocarcinoma, the functional significance of ROS dysregulation in solid tumors remain largely unstudied. The investigators aims are: (1) To characterize the frequency of ROS gene fusion, ROS protein overexpression and ROS gene mutations in cell lines and tumors from patients with hepatocellular carcinoma, colorectal, gastric, breast, ovarian, cholangiocarcinoma and non-small cell lung cancer, (2) To identify novel ROS gene variants in human solid tumors harboring ROS aberrations using next generation sequencing (NGS), (3) To determine the functional relevance of novel ROS gene variants identified with NGS, (4) To characterize the sensitivity of cells with functionally relevant ROS aberrations using ROS tyrosine kinase inhibitors. ROS fusions and protein overexpression will be screened in a panel of cell lines and primary tumors using Fluorescence In-situ Hybridization and immunohistochemistry respectively. Targeted next-generation sequencing will be applied to identify ROS variants in matching cancer types demonstrating high levels of gene fusion and protein overexpression. Functional characterization of novel ROS variants will be performed by silencing (shRNA) and overexpressing candidate cell lines with the respective ROS mutations/fusions, and evaluating their effects on biological functions including cell proliferation, migration, invasion and apoptosis, as well as sensitivity against ROS/ALK inhibitors. The investigators anticipate findings from this study will improve the investigators understanding of aberrant ROS signaling in an expanded group of cancer types, and potentially identifying a larger group of cancer patients that will benefit from ROS targeted therapy.

Further insight of the role of ROS receptor tyrosine kinase will confirm it as a therapeutic target in human solid tumors and hence expand the indication of crizotinib and other dual ALK/ ROS inhibitors. Furthermore, given the rarity of ROS fusion receptor tyrosine kinase in reported cancers, defining the epidemiology of ROS aberrations in other unreported cancers harboring ROS pathway activation is essential to properly design future clinical trials of ROS inhibitors. The validation of ROS receptor tyrosine kinase will also provide a new therapeutic target in the treatment of cancer and expand the role of novel targeted agents. Findings from this study will further the investigators knowledge on the oncogenic functions of the ROS and the application of ROS inhibitors in an extended group of solid tumors.

ELIGIBILITY:
Inclusion Criteria:

- Patients with cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Pathology, NUH Tissue Repository, The samples collected for the study are leftover clinical samples and the patients have consented for their samples to be used for research.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Characterize the frequency of ROS gene fusion, ROS protein overexpression and ROS gene mutations in cell lines and tumors
  To characterize the frequency of ROS gene fusion, ROS protein overexpression and ROS gene mutations in cell lines and tumors from patients with hepatocellular carcinoma, colorectal, gastric, breast, ovarian, cholangiocarcinoma and non-small cell lung cancer

SECONDARY OUTCOMES:
Identify novel ROS gene variants in human solid tumors harboring ROS aberrations using next generation sequencing (NGS)
Determine the functional relevance of novel ROS gene variants identified with NGS
Characterize the sensitivity of cells with functionally relevant ROS aberrations using ROS tyrosine kinase inhibitors

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore